CLINICAL TRIAL: NCT02637830
Title: In Situ Remineralisation Response of Different Artificial Caries-like Enamel Lesions to Home-care and Professional Fluoride Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Carolina Magalhães, Prof. Dr., University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 036/2011
Record Dates: First submitted 2015-12-08; First posted 2015-12-22 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — sodium fluoride topical preparation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Fluoride varnish and fluoride toothpaste (Experimental): Application of fluoride varnish (Duraphat) at the begining of the study. Application of fluoride toothpaste (Crest) twice a day for 3 days.
  Interventions: Other: Application of fluoride varnish (22600 ppm F, Duraphat) at the begining of the study; Other: Application of fluoride toothpaste (1500 ppm F, Crest) twice a day for 3 days of the study
- placebo toothpaste (Placebo Comparator): Application of placebo toothpaste twice a day for 3 days
  Interventions: Other: Application of placebo toothpaste (0 ppm F, Ice Fresh) twice a day for 3 days of the study
- Fluoride toothpaste (Active Comparator): Application of fluoride toothpaste (Crest) twice a day for 3 days
  Interventions: Other: Application of fluoride toothpaste (1500 ppm F, Crest) twice a day for 3 days of the study

INTERVENTIONS:
Other: Application of fluoride varnish (22600 ppm F, Duraphat) at the begining of the study
  Arms: Fluoride varnish and fluoride toothpaste
Other: Application of fluoride toothpaste (1500 ppm F, Crest) twice a day for 3 days of the study
  Arms: Fluoride toothpaste; Fluoride varnish and fluoride toothpaste
Other: Application of placebo toothpaste (0 ppm F, Ice Fresh) twice a day for 3 days of the study
  Arms: placebo toothpaste

SUMMARY:
This study mainly compared the response of the artificial carious enamel lesions to remineralisation in situ. The tested in vitro demineralising protocols were: MC gel, PA gel, MHDP and Buffer solutions.

The lesions were then remineralised in an in situ model, with crossover and double blind design. Fifteen volunteers wore intra-oral appliances containing 2 bovine enamel samples of each demineralising protocol during 3 experimental phases (3 days each). The experimental phases/treatments were: Control (Placebo dentifrice, saliva effect only), Home-care (fluoride dentifrice, 1,100 ppm F, NaF), and Professional/Home-care (varnish- 22,600 ppm F and dentifrice- 1,100 ppm F, NaF).

During the 3-day phase, the appliance was only removed during the main meals (four times a day, maximum 1 h duration each, interval between meals 2-3 h). Immediately after the meals, before replacing the appliance in the mouth, the subjects were advised to perform oral hygiene using a soft end-rounded toothbrush (Colgate® 360º Sensitive Pro-Relief TM) and dentifrice (non-fluoridated from IceFresh, Bauru, SP, Brazil or fluoridated dentifrice from Crest Procter & Gamble, Cincinnati, OH, USA) according to the phase and dental floss (Sanifill, São Paulo, Brazil).

The remineralising treatment with dentifrices was done ex vivo, 1 min twice a day (after the first and last oral hygiene of the day) using slurry of the dentifrice (1:3 water, 1 drop of solution/specimen). Thereafter, the appliance was replaced in the mouth and the subjects were advised to rinse with 10 ml of water for 5 s and to expectorate. In respect to Professional/Home-care phase, the varnish (Duraphat, Colgate, SP, Brazil) was applied before the in situ study for 6h and then removed.

The enamel remineralization was quantified using transverse microradiography (% mineral recovery and lesion depth, TMR), surface and cross-sectional hardness. The data were submitted to statistical analysis (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* a stimulated physiological salivary flow rate of >1 ml.min-1
* a non-stimulated physiological salivary flow rate of >0.25 ml.min-1
* good oral health (i.e. no cavities or significant gingivitis/periodontitis)

Exclusion Criteria:

* systemic illness
* pregnancy or breastfeeding
* use of fixed or removable orthodontic appliances
* use of fluoride mouthrinse or professional fluoride application in the last 2 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The increase of mineral content (% mineral volume) using transverse microradiography | 3 days
The increase of hardness (KHN or KgF/mm2) artificial caries lesions using surface and cross-sectional hardness | 3 days
Decrease of lesion depth (microns) of artificial caries lesions using transverse microradiography | 3 days